CLINICAL TRIAL: NCT06358196
Title: Complex Exploratory Study of Alcohol-Associated Hepatitis
Acronym: CESAH
Status: Not yet recruiting | Type: Observational
Sponsor: Pavol Jozef Safarik University (Other)
Collaborators: L Pasteur University Hospital (Unknown); Hospital Agel Kosice-Saca (Unknown); Technical University in Kosice (Unknown); Western University (Other); University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Jakub Gazda, Principial Investigator, Pavol Jozef Safarik University
Other Study IDs: CESAH
Record Dates: First submitted 2024-03-28; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Alcoholic Hepatitis
Keywords: alcoholic hepatitis; prognosis; epidemiology; treatment; hypothalamus-hypopituitary-adrenal axis; gut-Liver Microbiome Axis; nutritional status
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alcohol-associated hepatitis patients: Inclusion criterion
  • Patients older than 18 years with acute liver injury / acute liver failure with later confirmation of the AH diagnosis according to the NIAAA diagnostic criteria [14] who provided written informed consents for admission and further differentiation, and for study participation
  Exclusion criteria
  * Patients not confirmed to have alcohol-associated hepatitis
  * Patients with malignancies (specifically those with life-expectancy limitation)
  * Patients who withdrew consent for study participation

SUMMARY:
Alcohol-associated hepatitis is a clinical syndrome distinct from steatohepatitis or liver cirrhosis. It is associated with high mortality and characterized by an absence of effective treatment, while corticosteroids, which are currently used as the first-line treatment are effective only in a subpopulation of patients and only on 28-days survival - their effect on survival does not last beyond this interval. The proposed study is a complex exploratory study of alcohol-associated hepatitis with several epidemiology- and prognosis-related aims.

DETAILED DESCRIPTION:
Alcohol-associated hepatitis is a clinical syndrome distinct from steatohepatitis or liver cirrhosis. It is associated with high mortality and characterized by an absence of effective treatment, while corticosteroids, which are currently used as the first-line treatment are effective only in a subpopulation of patients and only on 28-days survival - their effect on survival does not last beyond this interval. The proposed study is a complex exploratory study of alcohol-associated hepatitis with the following aims: (1) to estimate the standardized annual incidence of (severe) AH in the Kosice Urban Area, (2) to estimate the threshold of alcohol consumption associated with (an increased risk of) developing AH, (3) to compare the diagnostic accuracy of NIAAA vs NIAAAm-CRP against liver biopsy, (4) to perform a head-to-head comparison of widely-accepted prognostic models and to develop prognostic models, (5) to observe prognosis of nonsevere alcohol-associated hepatitis, (6) to observe the evolution of severe alcohol-associated hepatitis, (7) to describe the association of hypothalamus-hypopituitary-adrenal axis and Gut-Liver Microbiome Axis and Prognosis of Alcohol-associated Hepatitis, (8) to describe the adherence to outpatient psychiatric management and its impact on long-term prognosis, (9) to perform a longitudinal evaluation of nutritional status, its changes, and its impact on long-term prognosis.

Study Design This is a multicenter observational study of patients with alcohol-associated hepatitis. The total trial duration for each subject is approximately 53 weeks. This includes a screening period of a maximum of one week (7 days), during which the diagnosis of AH will be confirmed, followed by a 52 weeks (365 days) observational period.

Diagnosis of Alcohol-associated Hepatitis The diagnosis of alcohol-associated hepatitis will be established using the National Institute on Alcohol Abuse and Alcoholism (NIAAA) diagnostic criteria: onset of jaundice within prior 8 weeks; ongoing consumption of >40 (females) or >60 (males) g alcohol/day ≥ 6 months, with less than 60 days of abstinence before the onset of jaundice; aspartate aminotransferase >0.83µkat/L (but less than 6.64 µkat/L), AST/ALT > 1.5, and total serum bilirubin > 51.3 mmol/L.

NIAAA definitions for AH differentiate between possible AH (clinically diagnosed with potential confounding factors), in which transjugular liver biopsy is indicated, probable AH (clinically diagnosed without potential confounding factors), and definite AH (clinically diagnosed and biopsy proven).

Considerations Regarding Patient Admission and Discharge Local standards dictate that patients with acute liver injury or acute liver failure are typically admitted to the 2nd Department of Internal Medicine, which specializes in gastroenterology and hepatology. This admission is carried out to facilitate further differentiation and provide specific treatment tailored to their condition. However, patients have the option to decline admission and, in such cases, will be discharged and managed as outpatients.

Once patients provide their consent to participate in the study, the screening period will commence. This screening phase may have a variable duration and will persist until a definitive diagnosis of AH is confirmed (either with or without results from histopathological evaluation of liver specimen).

The observational period will begin as soon as the diagnosis of AH will be confirmed with specific treatment in cases of sAH.

Patients diagnosed with nAH will undergo evaluation for potential discharge starting on Day 4 of the observational period. In contrast, patients with sAH will be assessed for their therapeutic response, as well as for the possibility of discharge, using the Lille score on Day 7 of the observational period. If patients do not respond to treatment, it will be discontinued.

For patients who respond positively to treatment, it will be sustained until Day 28 of the observational period. Following this period, treatment will be gradually tapered down by reducing the dosage by half each week, continuing for a total of three weeks.

The decision to discharge patients will be based on the absence of significant complications or serious events, such as gastrointestinal bleeding, overt hepatic encephalopathy, infection, kidney injury, and similar conditions. Similarly, if any of these events occur after discharge, patients will be promptly readmitted and receive appropriate treatment.

Patients will be offered psychiatric inpatient or outpatient care before discharge.

ELIGIBILITY:
Inclusion Criteria:

• Patients older than 18 years with acute liver injury / acute liver failure with later confirmation of the AH diagnosis according to the NIAAA diagnostic criteria [14] who provided written informed consents for admission and further differentiation, and for study participation

Exclusion Criteria:

* Patients not confirmed to have alcohol-associated hepatitis
* Patients with malignancies (specifically those with life-expectancy limitation)
* Patients who withdrew consent for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Alcohol-Associated Hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Standardized annual incidence of (severe) alcoholic hepatitis in the Kosice Urban Area | 1 year
  Number of patients with (severe) alcoholic hepatitis

SECONDARY OUTCOMES:
Threshold of alcohol consumption associated with (an increased risk of) developing AH | Baseline
  Grams of alcohol per week
Diagnostic accuracy of NIAAA and NIAAAm-CRP | Baseline
  Accuracy against liver biopsy
Prognostic performance of Maddrey, MELD, MELD-Na, MELD 3.0, GAHS, ABIC, Lille score | Baseline, Days 2, 4, 7
  Discriminatory characteristics (area under receiver operating characteristics curve) and calibration (calibration belts) with respect to 30 and 90 days mortality
Prognostic performance of SOFA and CLIF-C | Baseline, Days 2, 4, 7
  Discriminatory characteristics (area under receiver operating characteristics curve) and calibration (calibration belts) with respect to 30 and 90 days mortality
An update of Maddrey, MELD, MELD-Na, MELD 3.0, GAHS, ABIC, Lille score | Baseline
  To reevaluate independent variables in prognostic models aiming for improved discriminatory characteristics (area under receiver operating characteristics curve) and calibration (calibration belts)
Alternative to Lille model | Baseline, Day 2
  Regression model with 30 day mortality as exploratory variable
Prognostic model for 90 day survival | Baseline
  Regression model with 90 day mortality as exploratory variable
Uper limit of MELD or Maddrey scores beyond which patients no longer derive any therapeutic benefit from corticosteroid treatment | Baseline
  Upper threshold value of MELD and Maddrey scores associated with increased risk of mortality
Natural course of nonsevere alcoholic hepatitis | 1 year
  Mortality (and prevalence of ascites, hepatic encephalopathy, variceal bleeding, bacterial infection, acute kidney injury and proportion of patients with progression to severe alcoholic hepatitis)
Natural course of severe alcoholic hepatitis | 1 year
  Mortality (and prevalence of ascites, hepatic encephalopathy, variceal bleeding, bacterial infection, acute kidney injury and proportion of patients with progression to severe alcoholic hepatitis or with withdrawal syndrome, or with relapse of alcohol drinking)
Risk score for bacterial infection before corticosteroid treatment in patients with alcoholic hepatitis | Baseline
  30-days regression model for infection as exploratory variable
Distinguishing sterile Inflammation from infection in alcoholic hepatitis | 1 year
  Ratio of inflammatory markers
GUT microbiome and treatment response in alcoholic hepatitis | Baseline, Day 90
  Differences in GUT microbiome between corticosteroid responders and nonresponders
Hypothalamus-pituitary-adrenal axis and treatment response in alcoholic hepatitis | Baseline, Day 28
  Differences in cortisol levels between corticosteroid responders and nonresponders
Adherence to outpatient psychiatric management | 1 year
  Proportion of patients adhering to outpatient psychiatric management
Nutritional status and treatment response in alcoholic hepatitis | Baseline
  Differences in nutritional status between corticosteroid responders and nonresponders

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Gazda, MD, PhD, Principal Investigator — Pavol Jozef Safarik University
Locations (1):
- Pavol Jozef Safarik University, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No